CLINICAL TRIAL: NCT02549248
Title: Nanoparticles Analysis in Lung and Bronchi During Various Pulmonary Interstitial Diseases and Relationships With Their Aetiology. A Monocentric Study
Brief Title: Nanoparticles Analysis in Lung and Bronchi During Various Pulmonary Interstitial Diseases and Relationships With Their Aetiology
Acronym: NANOPI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1008122
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Interstitial Lung Diseases
Keywords: Interstitial Lung Diseases; nanoparticles; lung; broncho-alveolar lavage; bronchial washings
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavages (BAL), bronchial washings (BW), exhaled air condensates (EAC), blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiopathic interstitial diseases: " Test group ": patients suffering from idiopathic interstitial lung diseases including sarcoidosis and idiopathic pulmonary fibrosis.
  Nanoparticles (NP) loads will be measured on Bronchoalveolar lavages (BAL), bronchial washings (BW), exhaled air condensates (EAC), blood specimen and urine specimen.
  Interventions: Other: BAL; Other: BW; Other: EAC; Other: blood specimen; Other: Urine specimen
- Non idiopathic intertitial diseases: " Control group ": patients suffering from interstitial lung diseases of known aetiologies, such as hypersensibility pneumonitis, infectious or cancerous interstitial diseases and interstitial diseases caused by drug reactions.
  Nanoparticles (NP) loads will be measured on Bronchoalveolar lavages (BAL), bronchial washings (BW), exhaled air condensates (EAC), blood specimen and urine specimen.
  Interventions: Other: BAL; Other: BW; Other: EAC; Other: blood specimen; Other: Urine specimen

INTERVENTIONS:
Other: BAL — Patients with idiopathic and non idiopathic interstitial lung diseases
Other: BW — Patients with idiopathic and non idiopathic interstitial lung diseases
Other: EAC — Patients with idiopathic and non idiopathic interstitial lung diseases
Other: blood specimen — Patients with idiopathic and non idiopathic interstitial lung diseases
Other: Urine specimen — Patients with idiopathic and non idiopathic interstitial lung diseases

SUMMARY:
Nanoparticles (NP) are particles whose length, width and height are less than 100 nanometres. Over the past decade, industrial applications of NP have increased dramatically. Despite their widespread use, their true impact on human health remains unknown and poorly studied. NP exposure in humans primarily occurs via inhalation through the respiratory system. The aim of this study is to estimate the relationships between the nanoparticle load in the lung and bronchi and some interstitial lung diseases. In the aftermath of human exposure to asbestos, the pathological consequences of environmental exposure to nanomaterials could be evaluated upon a mineralogical analysis of pulmonary samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an interstitial lung disease assessed on clinical signs and CT scan, requiring a flexible bronchoscopy with a broncho-alveolar lavage.

These patients suffer from:

* Idiopathic interstitial lung diseases such as idiopathic pulmonary fibrosis or sarcoidosis OR
* Interstitial lung diseases of known aetiologies such as hypersensibility pneumonitis, infectious or cancerous interstitial diseases and interstitial diseases caused by drug reactions.

Written consent

Exclusion Criteria:

* Flexible bronchoscopy or BAL not possible.
* Pregnant women
* Patients under legal protection.
* Patients with contagious disease (HIV infection, tuberculosis, viral hepatitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * " Test group ": patients suffering from idiopathic interstitial lung diseases including sarcoidosis and idiopathic pulmonary fibrosis.
  * " Control group ": patients suffering from interstitial lung diseases of known aetiologies, such as hypersensibility pneumonitis, infectious or cancerous interstitial diseases and interstitial diseases caused by drug reactions.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
NP load | day 1
  The load of NP is a composite outcome. It will be described according to their level of presence (high, moderate or low), their size and chemical analysis.
  Analysis: The presence of NP will be assessed by dynamic light scattering (DLS). The elemental compositions of both the particulate (pellet) and the soluble (supernatant) fractions of each sample will be measured by means of inductively coupled plasma optical emission spectroscopy (ICP-OES). The samples for which DLS and ICP-OES corroborated a relatively stronger NP load will be observed under transmission electron microscopy (TEM) and field-emission electron microscopy (FESEM).

SECONDARY OUTCOMES:
Correlation between NP load in the lung and observed lung interstitial diseases | Day 1
  The load of NP is a composite outcome. It will be described according to their level of presence (high, moderate or low), their size and chemical analysis.
  The accurate diagnosis of the disease will be determined in accordance to the latest international guidelines, including the past history of each patient, the
  professional courses with focus on potential NP exposure, environmental studies, tobacco or drug use and exhaustive research of collagen or vascular diseases.
Correlation between NP load in the lung and NP load in blood specimen | Day 1
  The load of NP is a composite outcome. It will be described according to their level of presence (high, moderate or low), their size and chemical analysis.
Correlation between NP load in the lung and NP load in urine specimen | Day 1
  The load of NP is a composite outcome. It will be described according to their level of presence (high, moderate or low), their size and chemical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel VERGNON, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Derived] Marie-Desvergne C, Dubosson M, Leclerc L, Campo C, Bitounis D, Forest V, Pourchez J, Cottier M, Vergnon JM, Tarantini A, Chamel-Mossuz V. Characterization of the elemental and particle load of patient exhaled breath condensate and comparison with pulmonary lavages. J Breath Res. 2022 Dec 15;17(1). doi: 10.1088/1752-7163/aca697. PMID 36541529
- [Derived] Forest V, Pourchez J, Pelissier C, Audignon Durand S, Vergnon JM, Fontana L. Relationship between Occupational Exposure to Airborne Nanoparticles, Nanoparticle Lung Burden and Lung Diseases. Toxics. 2021 Aug 30;9(9):204. doi: 10.3390/toxics9090204. PMID 34564355